CLINICAL TRIAL: NCT02266212
Title: The Implications of Tobacco Smoking on Acute Postoperative Pain: A Prospective Observational Study
Brief Title: A Study on Analgesia and Related Outcomes for Patients With Tabacco Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yuan-Yi Chia, anesthesia doctor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS101-016
Record Dates: First submitted 2014-09-10; First posted 2014-10-16 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Current Smokers; Past Smokers; Never Smokers

ARMS (3):
- Smoke (Active Comparator): Fagerstrom test for nicotine dependence
  Interventions: Procedure: 5 ml arterial blood
- Pain (Active Comparator): pain during post-operation Day1 to Day4
  Interventions: Procedure: 5 ml arterial blood
- Morphine (Active Comparator): Morphine consumption during post-operation Day1 to Day4
  Interventions: Procedure: 5 ml arterial blood

INTERVENTIONS:
Procedure: 5 ml arterial blood — A sample of 5 ml arterial blood will be withdraw to test the arterial blood oxygen saturation, CO2 content, carbon monoxide (CO) content and carboxyhemoglobin (COHg).

SUMMARY:
Numbers of postoperative PCA(Patient-Controlled Analgesia) related side effects among current, past and non smokers are determined by comparing and analyzing frequency distributions. To determine whether smokers require more post operative opiate analgesics than others. Multivariate analysis will be performed to identify the major and the minor factors predicting the use of postoperative pain therapy. Our previous related study showed that the smoker male patients consumed more analgesics than those without smoking, but the female group showed the similar findings. However, the case number, especially the female cases, is underpowered. Investigators hope to increase the case number to have a better statistical and clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective general surgery are assigned to current smokers（n=100） or past smokers（n=100） or never smokers（n=100） according to the questionnaires "Fagerstrom test for nicotine dependence" 1 day prior to the surgery.

Exclusion Criteria:

* the patients undergoing major thoracic cardiovascular surgery
* the patients with significant lung lesion
* the patients with conscious disturbance
* the patients with allergic history to morphine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fagerstrom test for nicotine dependence | Post-operation Day1 to Day4

SECONDARY OUTCOMES:
Differences in pain intensity between the three groups after postoperative analgesia. | Post-operation Day1 to Day4
  Patients will give a pain score from 0 to 10. 10 is the most painful score.

OTHER OUTCOMES:
Morphine consumption | Post-operation Day1 to Day4
  Differences in postoperative morphine consumption between the 3 groups
side effects | Post-operation Day1 to Day4
  site effects include dizzy, vomit, lethargic sleep and pruritus

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan